CLINICAL TRIAL: NCT07184229
Title: Motivational Interviewing-Based Family Planning Counseling and Its Effect on Attitudes and Intentions Toward Modern Contraceptive Use Among Women Using Traditional Contraceptive Methods
Brief Title: Effect of Motivational Counseling on the Intention to Use Modern Contraceptive Methods
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Çiğdem Erdemoğlu, Dr, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/9-19
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Contraception
Keywords: traditional contraceptive methods; family planning; motivational interviewing; women

STUDY DESIGN:
Intervention Model Description: The study will include a total of 120 women, consisting of two control groups and one intervention group, each with 40 participants. The intervention group will receive motivational interviewing-based family planning counseling, the control group 1 will receive standard family planning counseling, and the control group 2 will receive no intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Family planning (Active Comparator): Standard family planning counseling
  Interventions: Behavioral: standard family planning counseling.
- Control (No Intervention): No intervention
- Motivational Interviewing (Experimental): Motivational interviewing-based family planning counseling
  Interventions: Behavioral: motivational interviewing-based family planning counseling

INTERVENTIONS:
Behavioral: motivational interviewing-based family planning counseling — This intervention consists of motivational interviewing-based family planning counseling aimed at women currently using traditional contraceptive methods. The counseling sessions are designed to enhance participants' motivation and readiness to adopt modern contraceptive methods by addressing their concerns, increasing knowledge, and resolving ambivalence. The comparator group will receive only standard family planning counseling.
  Other Names: standard family planning counseling
  Arms: Motivational Interviewing
Behavioral: standard family planning counseling. — The comparator group will receive only standard family planning counseling.
  Arms: Family planning

SUMMARY:
This study aims to evaluate the effect of motivational interviewing-based family planning counseling on attitudes and intentions toward modern contraceptive methods among women currently using traditional contraceptive methods. Despite the widespread use of traditional methods in many regions, including Turkey, modern contraceptive methods remain underutilized, leading to increased unintended pregnancies and related health burdens. Motivational interviewing is a client-centered counseling approach that supports individuals in making informed health decisions. By providing tailored counseling, this study seeks to improve women's awareness and motivation to adopt effective modern contraceptive methods, ultimately enhancing reproductive health outcomes. The findings are expected to contribute valuable insights for healthcare providers to improve family planning services and support women's reproductive choices.

DETAILED DESCRIPTION:
The motivational interviewing process consisted of 5 stages with 8 participants per group. A pre-interview will be conducted, followed by the first session one week later. The remaining four sessions will be held at two-week intervals, for a total duration of 9 weeks. The first and last sessions lasted 60 minutes; the others about 45 minutes. The stages of the motivational interviews were planned as follows:

Initial Session: Purpose and process explained, participant experiences assessed, and pre-tests conducted.

Engagement: Explored feelings and experiences about traditional family planning methods.

Supporting Self-Efficacy: Evaluated knowledge and confidence in modern methods. Change Talk: Focused on motivation and awareness for switching to modern methods.

Planning and Maintenance: Concrete action plans created, barriers and coping strategies discussed, and post-tests administered at the end.

ELIGIBILITY:
Inclusion Criteria:

Women aged between 18 and 49 years

* Literate in Turkish
* Currently using a traditional family planning method (e.g., withdrawal method)

Exclusion Criteria:

* Diagnosed psychiatric disorder
* Currently pregnant

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-16 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in attitude toward modern contraceptive methods | Before the intervention and 9 weeks post-intervention
  Assessed using a validated scale measuring women's attitudes toward modern contraceptive methods.
  Family Planning Attitude Scale: The scale was developed by Örsal and Kubilay in 2007. It is a 5-point Likert-type scale consisting of 34 items. Each statement on the scale is scored as "1=Strongly Agree," "2=Agree," "3=Undecided," "4=Disagree," and "5=Strongly Disagree." The scale has three subdimensions: attitudes toward family planning in society (items 1-15), attitudes toward family planning methods (items 16-26), and attitudes toward childbirth (items 27-34). The attitude toward family planning in society subdimension scores range from 15 to 75, the attitude toward family planning methods subdimension scores range from 11 to 55, the attitude toward childbirth subdimension scores range from 8 to 40, and the total scale score ranges from 34 to 170. As the score on the scale increases, the attitude toward family planning becomes more positive.

SECONDARY OUTCOMES:
Change in intention toward modern contraceptive methods | Before the intervention and 9 weeks post-intervention
  Assessed using a validated scale measuring women's intention toward modern contraceptive methods.
  The Contraceptive Intention Scale (CIS) was developed by Bennet and Rocca in 2015 to assess contraceptive intention.12 The Turkish validity and reliability study of the scale was conducted by Suid and Pasinlioğlu in 2016.19 The scale consists of a total of 15 items and uses a 4-point Likert-type format. The minimum possible total score on the scale is 0, and the maximum is 15. An increase in the score indicates a higher contraceptive intention.

CONTACTS AND LOCATIONS:
Locations (1):
- K-8 Containerkent, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Demographic data and survey results, with all personal identifiers removed, will be shared with researchers at the time of publication.
Time Frame: IPD will be available starting 6 months after publication and will remain accessible for 3 years.
Access Criteria: Access will be granted to qualified researchers upon reasonable request and after approval by an independent review committee.